CLINICAL TRIAL: NCT07219121
Title: A Multicenter, Open-label Single Arm Study to Evaluate the Safety and Efficacy of Sparsentan in Posttransplant Immunoglobulin A Nephropathy (IgAN) or Focal Segmental Glomerulosclerosis (FSGS) (SPARX)
Brief Title: Sparsentan in Posttransplant Immunoglobulin A Nephropathy or Focal Segmental Glomerulosclerosis
Acronym: SPARX
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Travere Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TVTX-RE021-426
Record Dates: First submitted 2025-10-09; First posted 2025-10-21 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Proteinuria; Immunoglobulin A (IgA) Nephropathy; Focal Segmental Glomerulosclerosis; Kidney Transplant
Keywords: IgAN; FSGS; kidney transplant; proteinuria
MeSH Terms: conditions — Proteinuria; Kidney Diseases; Glomerulosclerosis, Focal Segmental | interventions — sparsentan

STUDY DESIGN:
Intervention Model Description: 46-week, open-label, multicenter, single-group Phase 4 study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Drug: Sparsentan (Experimental): A non-immunosuppressive single molecule with dual antagonism of ETAR and AT1R, has shown potent anti-proteinuric effect in patients with native kidney disease, including IgAN and FSGS.
  Interventions: Drug: Sparsentan

INTERVENTIONS:
Drug: Sparsentan — For participants with a kidney transplant with IgAN:
  Day 1 through Week 2 visit, participants will take 200 mg once daily (QD) prior to the morning meal. At the Week 2 visit, participants will titrate up to 400 mg QD and take this dose through Week 36, if tolerated and determined to be safe by the Investigator.
  For participants with a kidney transplant with FSGS, or a biopsy finding of both IgAN and glomeruli with FSGS patterns:
  Day 1 through Week 2 visit, participants will take 400 mg QD prior to the morning meal. At the Week 2 visit, participants will titrate up to 800 mg QD and take this dose through Week 36, if tolerated and determined to be safe by the Investigator.

SUMMARY:
To evaluate the safety and efficacy of sparsentan tablets for the treatment of patients with proteinuria after kidney transplantation with once-daily dosing for 36 weeks.

DETAILED DESCRIPTION:
This is a 46-week, open-label, multicenter, single-group Phase 4 study to determine the safety and efficacy of sparsentan for the treatment of patients post kidney transplantation with IgAN or FSGS with proteinuria (≥ 0.5 g/g).

Eligible participants with a kidney transplant receiving stable standard of care (SOC) therapy, including standard immunosuppressive therapy (IST) to prevent graft rejection, will be enrolled to receive sparsentan treatment for 36 weeks. Participants will remain on standard IST for the duration of the study and will stop RAASi prior to initiating sparsentan treatment. The final dose of a RAASi should be taken on the day before the Day 1 visit.

Participants with a kidney transplant, at least one year prior to screening, with biopsy-proven IgAN will take 200 mg orally once daily (QD) for 2 weeks, then 400 mg QD through Week 36. Participants with a kidney transplant with FSGS histological pattern in the graft, or a biopsy finding of both IgAN and glomeruli with FSGS patterns will take 400 mg orally QD for 2 weeks, then 800 mg QD through Week 36.

Study visits will be conducted at Day 5 and Weeks 2, 4, 6, 12, 24, and 36 following Day 1. Following the 36 week treatment period, all participants will complete a 4 week off-sparsentan treatment follow-up period (ie, no study drug), during which time treatment will be at the discretion of the investigator. Participants will have a telephone visit at Week 40.

ELIGIBILITY:
Inclusion Criteria:

* Willing and capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the ICF and in the protocol.
* Male and female aged ≥18 years
* Participants with a kidney transplant with biopsy-proven IgAN or FSGS histological pattern in the graft.
* A period of ≥12 months since kidney transplantation.
* UPCR ≥0.5 g/g and eGFR (CKD-EPI creatinine-based formula ≥30 mL/min/1.73 m2.
* Participants who can become pregnant, must agree to the use of 1 highly reliable method of contraception from 7 days prior to the first dose of study intervention until 30 days after the last dose of study intervention.
* Systolic BP ≤160 mmHg and ≥100 mmHg, and diastolic BP ≤100 mmHg and ≥60 mmHg at screening.
* For participants on an ACEI and/or ARB, and/or sodium glucose cotransporter-2 (SGLT2) inhibitor, the dosing regimen(s) is stable for ≥6 weeks prior to screening.

Exclusion Criteria:

* Participant has multiorgan transplants (with the exception of pancreas and corneal transplants).
* Immunosuppressive therapy (IST) regimen for kidney transplant or other systemic chronic ISTs including enteric budesonide that is not stable for >6 weeks prior to Day 1. Exceptions include routine changes in the dose of CNIs to meet target level.
* <3 months after antirejection treatment and active rejection.
* Active bacterial, fungal or viral infection and/or active treatment of infection including BK virus (BKV), cytomegalovirus (CMV), human immunodeficiency virus (HIV), Hepatitis B and C <3 months prior to and during the screening period.
* Current treatment for surgical complications.
* History of heart failure (New York Heart Association [NYHA] Class II-IV).
* Jaundice, hepatitis, or known hepatobiliary disease.
* Malignancy within the past 2 years with the exception of adequately treated basal cell carcinoma or non-metastatic squamous cell carcinoma of the skin, with no evidence or recurrence.
* History of alcohol or illicit drug use disorder (as defined in the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition).
* History of serious side effects or allergic response to any angiotensin II antagonist or ERA.
* Participant requires any of the prohibited concomitant medications.
* Treatment with sparsentan <12 weeks prior to screening.
* Participant has participated in a study of another investigational product <28 days prior to screening or plans to participate in such a study during the course of this study.
* Hematocrit <27%, hemoglobin <90 g/L (9 g/dL), or potassium >5.5 mmol/L (5.5 mEq/L).
* The participant is pregnant, plans to become pregnant during the course of the study, or is breastfeeding.
* The participant, in the opinion of the Investigator, is unable to adhere to the requirements of the study, including the ability to swallow the study IMP whole.
* The participant, in the opinion of the Investigator, has a medical condition or abnormal clinically significant laboratory screening value not listed above that may interfere with the evaluation of sparsentan safety or activity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-10-07 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Urinary protein/creatinine ratio (UPCR) | 36 weeks
  Change from baseline (Day 1) in urinary protein/creatinine ratio (UPCR) to Week 36.

SECONDARY OUTCOMES:
Change from baseline in UPCR | 36 weeks
  Change from baseline in UPCR each visit.
Urinary albumin/creatinine ratio (UACR) | 36 weeks
  Change from baseline in UACR at each visit
Change from baseline in eGFR (estimated glomerular filtration rate) | 36 weeks
  Change from baseline in eGFR, applying creatinine and cystatin C based formulae, at each visit
Change from baseline in blood pressure (BP) | 36 weeks
  Change in systolic and diastolic BP at each visit
Achievement of UPCR <0.3 g/g | 36 weeks
  Achievement of UPCR <0.3 g/g at Weeks 12, 24 and 36
30% and 50% reductions in UPCR | 36 weeks
  The proportion of participants achieving 30% and 50% reductions in UPCR at Week 36.

CONTACTS AND LOCATIONS:
Overall Officials: Radko Komers, MD, PhD, Study Director — Travere Therapeutics
Locations (9):
- United States (9):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Cornell Medical Center, New York, New York
  - University of North Carolina Chapel Hill, Mooresville, North Carolina
  - Ohio State University, Columbus, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Dallas Nephrology Associates, Dallas, Texas
  - University of Texas, Galveston, Texas
  - University of Washington, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Requests for clinical trial data, including language stating its intended use, should be directed to datarequest@travere.com. If approved, the requested information will be provided to the requestor after signing a data access agreement. Requests can be made following completion of the study and full publication of the study data in a peer reviewed journal for up to 36 months following its publication. Travere reserves the right to decline or recommend modifications to a request if it does not comply with the data sharing policy or if it is determined that the request is made by a biased source.
Time Frame: Requests can be made following completion of the study and full publication of the study data in a peer reviewed journal for up to 36 months following its publication.